CLINICAL TRIAL: NCT02305173
Title: Effect of the Preoperative Administration of Dexamethasone in the Respiratory Function and Postoperative Symptoms in Women Undergoing Mastectomy for Cancer. Results of a Randomized Clinical Trial.
Brief Title: Dexamethasone and Respiratory Function After Mastectomy
Acronym: Dexa-mama
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, GONZALEZ-OJEDA ALEJANDRO, Alejandro González-Ojeda, Ph.D., M.D., Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Dexamethasone-2014-4
Record Dates: First submitted 2014-11-20; First posted 2014-12-02 (Estimated); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Respiratory; Disorder, Functional, Impaired
Keywords: dexamethasone; pulmonary function; spirometry; mastectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dexamethasone group (Active Comparator): patients receive one single dose of intravenous dexamethasone 8 mg.
  Interventions: Drug: Intravenous Dexamethasone
- placebo group (Placebo Comparator): patients receive one single dose of intravenous placebo.
  Interventions: Drug: intravenous salin water

INTERVENTIONS:
Drug: Intravenous Dexamethasone — One dose of intravenous dexamethasone (8 mg) 60 minutes before surgery.
  Other Names: no other intervention
  Arms: dexamethasone group
Drug: intravenous salin water — Patients of the control group received homologated placebo 60 minutes before surgery.
  Other Names: no other intervention
  Arms: placebo group

SUMMARY:
Preoperative dexamethasone reduces symptoms after different surgical procedures including mastectomy in breast cancer, but the effect in the postoperative respiratory function remains unknown. The aim of this protocol was to determine if the administration of a single dose of dexamethasone during the preoperative, could improve respiratory function and postoperative symptoms of patients undergoing mastectomy in breast cancer.

DETAILED DESCRIPTION:
Controlled clinical trial will be performed in 120 surgical patients treated for breast cancer, conducted from Nov 2014 to Nov 2015. Patients will be divided in three groups: Group 1 consisted in patients who underwent conservative breast with axillary lymph node dissection, group 2 in patients with radical mastectomy without reconstruction, and group 3 patients with radical mastectomy with immediate reconstruction with synthetic breast implants.

All patients will be randomly assigned by a system of sealed envelopes, to receive 8 mg of intravenous dexamethasone or placebo 60 minutes before surgery. All patients will be female and had a confirmed diagnosis of breast carcinoma. The investigators will exclude patients with a classification of the American Society of Anesthesiologists classes III and IV. Other exclusion criteria are: age 80 years, pregnancy or during menstruation, during steroid therapy, severe diabetes mellitus (serum HbA1c> 8%); opioids, sedatives or painkillers less than a week before the mastectomy, or a history of alcohol or drugs. The investigators will exclude patients with a history of inner ear disease and / or severe PONV after any surgical procedure performed in the past. All patients will be admitted to hospital one day before surgery and were followed from hospital admission and until 30 days after surgery for any medical or surgical morbidity.

Anesthesia and surgery

All patients will be standardized to the next anesthetic protocol:

Under venipuncture, patients receive 1 g of Cephalothin IV one hour before starting the procedure. After entering the operating room, type 1 continuous monitoring was placed via noninvasive, Midazolam will be administered via peripheral 0.1-0.2 mg/kg as well as fentanyl 1 mcg / kg IV. Prongs will be placed and basal hemodynamic values will be taken with preoxygenation by tidal volume technique per minute.

Induction will be performed with Propofol 1-2 mg/kg IV and completed with fentanyl (3 mcg / kg IV) along with the administration of Rocuronium 0.06 mg/kg IV. Assisted oxygenation continues at a rate of 5 lpm and laryngeal mask (mask measure according to weight and body distribution of the patient) is placed.

During surgery, the medication will be completed with omeprazole 40 mg IV, Ondancetron 4 mg IV. All patients will be monitored with indirect determinations of blood pressure and heart rate using standard techniques, as well as the content of expired CO2 and oxygen saturation of the blood. Subsequently, all patients will be extubated and transferred to the unit for immediate post-surgical care with cardiovascular monitoring and oxygen.

Surgical Procedures All patients will be submitted to treatment according to the clinical stage with conservative breast surgery with axillary dissection, radical mastectomy without immediate reconstruction or radical mastectomy with immediate reconstruction with synthetic implants. In case of radical mastectomy, a closed drainage system will be placed in the chirurgic region, and will be removed when drainage is less than 50ml in 24 hours. Chemotherapy or radiation therapy will be administered 3-4 weeks following surgical resection.

Analgesic and antiemetic therapy Nonsteroidal antiinflammatory drugs will be used as analgesia after surgery with sodium ketorolac 30 mg IV every 6 hours (in patients younger than 60 years) or lysine Clonixinate 100 mg IV every 6 hours (in patients older than 60 years). Also, patients who will be submitted to a conservative surgery will receive intravenous Tramadol 100mg (diluted in 50ml of solution); the dose may be repeated every 12 hours until. Repeated doses of Morphine of 2.5 mg IV will be used in case of radical mastectomy, according to the needs of the patient. If pain is not diminish within 30 minutes a VAS will be used and in case the scale is greater than 7, an infusion of 10mg of morphine in 250ml 0.9% of saline solution will be used. Pain will be assessed on return to the recovery room and at 6, 12 and 24 h postoperatively using a visual analogue scale (VAS; 0 = no pain and 10 = most severe pain).

The incidence of PONV will be recorded immediately on return to the recovery room and at 6, 12 and 24 h postoperatively using a three-point ordinal scale (0 = asymptomatic, 1 = feeling of nausea or tonnage without expulsion oral route of gastric contents 2 = vomiting). Nausea is defined as a unpleasant sensation associated with awareness of the urge to vomit; retching is defined as the labored, spasmodic rhythmic contraction of the respiratory muscles without the expulsion of gastric contents, and vomiting is defined as the forceful expulsion of gastric contents from the mouth. Ondancetron will be used IV (4-8 mg) to treat these symptoms.

Pulmonary Function. To perform a spirometry, the ambient must comply the following characteristics: environment without audio or visual shocks and thermal comfort for the comfort of the patient. Patients will be told to sit in a comfortable position with your back straight (at an angle greater than 45°, to patient tolerance) and high chin. Lightweight support will be perform in the patient by taking her gently by the shoulders to keep them lean forward and off balance grew. In the immediate postoperative and due to postoperative pain, the patient will be settled in the stretcher to emulate the sitting position (inclination greater than 45 °) performing the previously mentioned subject. The nature of the study will be explained in understandable language to the patient, and their cooperation will be requested. Forced espiratory maneuver will be explained and immediately exemplified by the best qualified to understand the patient and to avoid measurement bias evaluator. Special emphasis will be placed on the importance of starting the effort with the maximum volume of air in the lungs, so determined and energetic, as well as maintaining exhalation as long as possible. She will be asked to take the disposable cardboard mouthpiece adaptable to pneumotachograph, sealing it with the lips in the position of maximal inspiration and then blow air through it, initiating a sharp exhalation maneuver with the above characteristics. To be a valid test, the maneuver should be performed with a proper effort, starting from the position of maximal inspiration without hesitation or false start with a continuous exhalation without corrections, cough or Valsalva maneuver, as well as checking for leaks were recorded in nozzle. A total of three satisfactory maneuvers will be performed with a maximum of eight attempts for each measurement, spaced at least for 30 seconds. To perform the study, a "Fleisch spirometer" with brand Sibelmed® neumotac type model will be used Datospir 110/120.

Measurements of forced espiratory volume in one second (FEV1), forced vital capacity (FVC) Maximum Forced Espiratory Flow (FEFM) and the ratio between forced espiratory volume in one second and forced vital capacity will be taken into account (FEV1 / FVC). Such clinical parameters are directly related to muscle fatigue, the compliance of the lung parenchyma and respiratory status of patients.

Statistical Analysis Postoperative complications will be recorded during hospitalization and patients will be followed up to 30 days after hospital discharge. Data collected will include patient age, body mass index (BMI), smoking history and neoadjuvant chemotherapy, anesthesia and operation time and the frequency of use of analgesics and antiemetics. These parameters will be added and compared between dexamethasone and placebo groups. The endpoints of the study will be postoperative nausea and vomiting, and pain measured by the VAS and the need for additional analgesia and antiemetic drugs as described.

The sample size was predetermined. The investigators expect a 35% difference in the incidence of nausea and vomiting between groups. The α error 0.05 and β error 0.20; n = 35 patients in each group will be considered adequate, according to an analysis of power. All results eill be expressed as percentages and means with standard deviation ± (SD). Student t test, Chi 2 of Fisher's exact test will be used to analyze quantitative and qualitative data, respectively. Differences will be considered statistically significant at p <0.05.

Ethical Considerations This protocol has been registered with the Local Research and Ethics Committee on Health.

The study will be conducted according to the principles of the Helsinki Declaration of 1989, and with the Guidelines of Health of Mexico. The local research and ethics committee of Health Research Ethics Committees of the Cancer Institute of Jalisco, Mexico approved all protocols. A full written informed consent will be obtained from all patients before inclusion in the study.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of breast carcinoma

Exclusion Criteria:

* patients with a classification of the American Society of Anesthesiologists classes III and IV.
* pregnancy
* during menstruation
* during steroid therapy
* severe diabetes mellitus (serum HbA1c> 8%)
* opioids, sedatives or painkillers less than a week before the mastectomy
* history of alcohol or drugs
* patients with a history of inner ear disease and / or severe PONV after any surgical procedure performed in the past

Ages: 20 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-11; Primary Completion 2015-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change in Forced Vital Capacity (FVC), measured in Liters/second and in percentage %. | change occurred from 1 hour before surgery and after 1, 6, 12 and 24 postoperative hours
  maximum amount of air a person can expel from the lungs after a maximum inhalation.
Change in Forced Espiratory Volume (FEV) in the first second, measured in Liters/second and in percentage %. | change occurred from 1 hour before surgery and after 1, 6, 12 and 24 postoperative hours
  Measures the amount of air a person can exhale during a forced breath in one second.
Change in Peak Respiratory Flow (PRF). measured in Liters/second and in percentage %. | change occurred from 1 hour before surgery and after 1, 6, 12 and 24 postoperative hours
  A person maximum speed of expiration

SECONDARY OUTCOMES:
Change in pain occurred from 1 hour before surgery and after 1, 6, 12 and 24 hours after surgery. | change occurred from 1 hour before surgery and after 1, 6, 12 and 24 postoperative hours
  An unpleasant sensation occurring in varying degrees of severity as a consequence of injury, disease, or emotional disorder.
Change in nausea occurred from 1 hour before surgery, and after 1, 6, 12 and 24 hours after surgery. | change occurred from 1 hour before surgery and after 1, 6, 12 and 24 postoperative hours
  Nausea is the feeling of having and urge to vomit. It is often called being sick to your stomach.
Change in vomiting occurred from 1 hour before surgery, and after 1, 6, 12 and 24 hours after surgery. | change occurred from 1 hour before surgery and after 1, 6, 12 and 24 postoperative hours
  Vomiting is forcing the contents of the stomach up through the esophagus and out of the mouth.
Total dose of backup analgesic medication administrated to each patient | 24 hours after surgery
  Total dose of backup analgesic medication will be recorded during the last 24 hours after the surgical procedure.
Total dose of backup antiemetic medication administrated to each patient | 24 hours after surgery
  Total dose of backup antiemetic medication will be recorded during the last 24 hours after the surgical procedure.
Morbidity after mastectomy | 24 postoperative hours and until 8 days after surgery after hospital discharge.
  The prevalence of a disease in a particular percentage of the population; the number of cases of a particular disease per unit of population.
Change in Oximetry (percentage %). | change occurred from 1 hour before surgery and after 1, 6, 12 and 24 postoperative hours
  Determination of the oxygen saturation of arterial blood using an oximeter.

CONTACTS AND LOCATIONS:
Overall Officials: González-Ojeda Alejandro, PhD. MD., Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Research Unit in Clinical Epidemiology, Specialties Hospital. Mexican Institute of Social Security, Guadalajara, Jalisco, Mexico

REFERENCES:
- [Derived] Jimenez-Tornero J, Cortes-Flores AO, Chavez-Tostado M, Morgan-Villela G, Zuloaga-Fernandez Del Valle C, Zuloaga-Fernandez Del Valle R, Garcia-Gonzalez LA, Fernandez-Avalos VS, Miranda-Ackerman RC, Alvarez-Villasenor AS, Ambriz-Gonzalez G, Barbosa-Camacho FJ, Fuentes-Orozco C, Contreras-Cordero VS, Gonzalez-Ojeda A. Effect of a preoperative single-dose steroid on pulmonary function and postoperative symptoms after modified radical mastectomy: results of a randomized clinical trial. Gland Surg. 2020 Oct;9(5):1313-1327. doi: 10.21037/gs-20-366. PMID 33224806